CLINICAL TRIAL: NCT00840385
Title: Phase II Study of Orally Fludarabine, Adriamycin and Dexamethasone (FAD) in Newly Diagnosed PTCL
Brief Title: Orally Fludarabine, Adriamycin and Dexamethasone (FAD) in Newly Diagnosed Peripheral T-cell Lymphomas (PTCL)
Acronym: FAD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Base for drug clinical trials, Fudan University cancer hospital, Fudan University cancer hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-71-143
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Last update posted 2010-09-15 (Estimated); Status verified 2010-09

CONDITIONS: T-Cell Lymphomas; Chemotherapy
Keywords: Peripheral T-cell lymphomas (PTCL); Fludarabine
MeSH Terms: conditions — Lymphoma, T-Cell; Lymphoma, T-Cell, Peripheral | interventions — Flavin-Adenine Dinucleotide; fludarabine phosphate; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: FAD

INTERVENTIONS:
Drug: FAD — Fludarabine 40mg/m2 po.d1-3; Adriamycin 50mg/m2 i.v.d1; Dexamethasone 20mg/d po.d1-5.
  Other Names: Fludarabine phosphate; oral fludarabine

SUMMARY:
The primary objective of this study is to evaluate the efficacy of Fludarabine, Adriamycin and Dexamethasone (FAD) as first line therapy in patients with Peripheral T-cell lymphomas (PTCL). 30 patients will be treated into this study.

DETAILED DESCRIPTION:
Doxorubicin is often used to treat Peripheral T-cell lymphomas (PTCL). However, patients with PTCL have an especially poor outcome with a 5-year overall survival rate of only 26% following treatment with standard doxorubicin containing regimens. There is general agreement that results with conventional chemotherapy are so poor in patients with most PTCL that new approaches are warranted.The nucleoside analogs are Fludarabine being combined with other agents in PTCL (excluding ALK positive ALCL and primary cutaneous ALCL) is reported by others.We conduct a II stage clinical trials to evaluate the efficacy of Orally Fludarabine, Adriamycin and Dexamethasone (FAD) as first line therapy in patients with in Newly Diagnosed PTCL.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of peripheral T cell lymphoma must established by histological biopsy, and immunochemistry analysis and cytogenetic assessment should be done as well. The patients with peripheral T cell lymphoma (PTCL), PTCL-unspecified type(PTCL-u), angioimmunoblastic lymphoma (AILT) and non-skin type anaplastic large cell lymphoma (ALCL, ALK-).
2. Aged 18~75.
3. Good performance status, ECOG score≤2. Estimated survival span >3 months
4. Previously untreated.
5. At least 1 assessable disease (maximal diameter >1.0cm, the disease foci located within the irradiated area are excluded) evaluated by CT or MRI, PET is also permitted.
6. Good compliance and inform consenting
7. Fit for the following criteria:

   * Absolute neutrophil count (ANC)≥1.5×109/L
   * Platelet（PLT）≥80×109/L
   * Total bilirubin (TBI) ≤upper normal limit (UNL)
   * Serum creatine (Cr) ≤UNL
   * Alanine aminotransferase (ALT) and Aspartate transaminase（AST）≤1.5 UNL

Exclusion Criteria:

1. Severe cardiac, renal or hepatic incompetence: serum direct bilirubin, indirect bilirubin, ALT, AST and Cr greater than 1.5 UNL; cardiac function greater than grade II. 28 days within the major surgical operation.
2. Other malignancy history (skin basement cell carcinoma and cervical carcinoma are excluded)
3. Severe uncontrolled underlying diseases
4. Pregnancy or lactation
5. Autoimmune disease history
6. Severe infection or metabolic diseases
7. Known allergic to multiple agents, including sulphanilamide.
8. Severe peptic ulceration or bleeding, contra-indicative for corticosteroids
9. Lymphoma involving central nervous system

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-11; Primary Completion 2010-11 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
side effects | 1 months

SECONDARY OUTCOMES:
PFS (progression free survival) | 3 months
complete remission(CR) | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiaonan Hong, MD, Principal Investigator — Fudan University
Locations (1):
- Cancer Hospital, Fudan University, Shanghai, Shanghai Municipality, China